CLINICAL TRIAL: NCT05565430
Title: Vocal Cord Responses During Hyperventilation in Normal Individuals and in Mild and Severe
Brief Title: Vocal Cord Responses During Hyperventilation in Normal Individuals and in Mild and Severe Asthmatics.
Status: Completed | Type: Observational
Sponsor: Monash Medical Centre (Other)
Responsible Party: Principal Investigator, Laurence Ruane, Respiratory Scientist, Monash Medical Centre
Other Study IDs: 16151A
Record Dates: First submitted 2016-05-31; First posted 2022-10-04 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-10

CONDITIONS: Hyperventilation; Larynx; Asthma
Keywords: Hyperventilation; Asthma; Vocal Cords; Extra-thoracic airway hyper-responsiveness; Anti-cholinergics
MeSH Terms: conditions — Hyperventilation; Laryngeal Diseases; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Control: 1. Acute Hyperventilation and effects on vocal cord movement.
  2. Chronic Hyperventilation and effects on vocal cord movement.
  3. Effects of anticholinergic medication on paradoxical vocal cord movement.
  Interventions: Other: Acute Hyperventilation; Other: Chronic hyperventilation; Drug: Effects of anticholinergic medication
- Mild Asthmatics: 1. Acute Hyperventilation and effects on vocal cord movement.
  2. Chronic Hyperventilation and effects on vocal cord movement.
  3. Effects of anticholinergic medication on paradoxical vocal cord movement.
  Interventions: Other: Acute Hyperventilation; Other: Chronic hyperventilation; Drug: Effects of anticholinergic medication
- Severe Asthmatics: 1. Acute Hyperventilation and effects on vocal cord movement.
  2. Chronic Hyperventilation and effects on vocal cord movement.
  3. Effects of anticholinergic medication on paradoxical vocal cord movement.
  Interventions: Other: Acute Hyperventilation; Other: Chronic hyperventilation; Drug: Effects of anticholinergic medication

INTERVENTIONS:
Other: Acute Hyperventilation — Laryngoscopy to assess vocal cord function during acute hyperventilation in normal subjects and asthmatics.
  Other Names: Acute Hyperventilation in normal subjects and asthmatics
Other: Chronic hyperventilation — Laryngoscopy to assess vocal cord function during acute hyperventilation in normal subjects and asthmatics.
Drug: Effects of anticholinergic medication — Laryngoscopy to assess vocal cord function after administration of anticholinergic medication.
  Other Names: Effects of anticholinergic medication on vocal cord movement

SUMMARY:
The Investigators aim to:

1. Study the effect of hyperventilation on the development of paradoxical vocal cord movement (PVCM) in healthy individuals and in patients with mild and severe asthma,
2. Relate PVCM to airway symptoms and measurements of intra- and extra-thoracic airway hyperresponsiveness (ET-AHR),
3. Evaluate the effects of inhaled anti-cholinergic agents on PVCM induced by hyperventilation.

Hypotheses:

1. In health PVCM will not occur in response to hyperventilation,
2. In asthma PVCM will occur in response to hyperventilation,
3. Airway symptoms and ET-AHR will develop in parallel with PVCM,
4. Inhaled anticholinergic agents will prevent PVCM induced by hyperventilation.

DETAILED DESCRIPTION:
Specific aims:

Project 1 - 'Acute' hyperventilation in normal subjects and asthmatics.

Aim 1.1: To measure PVCM by endoscopy in response to a single period of hyperventilation in normal subjects and asthmatics.

Aim 1.2: To relate PVCM to symptoms in both groups. Aim 1.3: To relate PVCM to bronchial and ET-AHR before and after acute hyperventilation.

Project 2 - 'Chronic' hyperventilation and the effect on vocal cord movements in asthmatic subjects.

Aim 2.1: To measure PVCM by endoscopy in response to multiple periods of hyperventilation (twice daily over 2 weeks) in normal subjects and asthmatics.

Aim2.2: To relate PVCM to symptoms in both groups. Aim 2.1: To relate PVCM to bronchial and ET-AHR before and after chronic hyperventilation.

Project 3 (a) - Effects of anticholinergic medication on PVCM.

Aim 3.1: Determine the effect of anti-cholinergic inhaled medications on PVCM induced by hyperventilation.

Project 3 (b) - PVCM during exercise and the effects of anticholinergic medication on PVCM If no PVCM is detected in project 1 and 2, as an alternative strategy the Investigators will examine PVCM that has been shown to occur in severe asthma in response to exercise. The effect of anti-cholinergic inhaled medications will then be examined in this model.

Significance:

Dysfunctional breathing may be a mechanism whereby symptomatic PVCM develops in asthma but not in health. The proposed studies will enhance the Investigators understanding of the role played by dysfunctional breathing in the pathogenesis of this distressing condition and may provide a rationale for targeted therapies.

ELIGIBILITY:
Inclusion Criteria for Healthy Controls:

* Inclusion criteria for healthy controls include:

  * age >18 to 65 years old
  * non-smokers
  * No history of chronic respiratory symptoms.

Exclusion Criteria for Healthy Controls:

* Exclusion criteria for controls include:

  * Age < 18 or > 65, smokers or smoking history >10 pack years
  * Any history of respiratory disorders such as asthma or chronic obstructive pulmonary disease (COPD)
  * Known vocal cord pathology (i.e. laryngeal cancer) or diagnosed voice condition
  * Known brain or brainstem cancer
  * Known head and neck cancer
  * Known neurological disorders (i.e. stroke)
  * Use of medications (i.e. beta-blockers or anti-cholinergic agents which may interfere with vocal cord function)
  * Singers
  * Pregnancy.

Inclusion Criterial for Asthmatics:

* The Investigators shall recruit a total of 16 patients with asthma - 8 patients with mild asthma (Group 2) and 8 patients with severe asthma (Group 3).

  * Mild asthma will be defined as patients with forced expiratory volume in 1 second (FEV1) >80% predicted.
  * Severe asthma will be defined as patients with FEV1 50-60% predicted.
  * Asthmatics will also have a forced expiratory ratio (FER) less than the lower limit of normal, indicating obstruction.
* Inclusion criteria will include:

  * age 18-65 years
  * A history of asthma defined as a bronchodilator response with increase in FEV1 >12% and 200mls or positive bronchoprovocation testing (methacholine).
  * Asthmatics will have FEV1 >50% predicted.

Exclusion Criteria for Asthmatics:

- Exclusion criteria will include:

* Age < 18 or > 65
* Smoking history > 10 pack years,
* FEV1 < 50% predicted
* Allergy to anti-cholinergics, known COPD
* Known vocal cord pathology (i.e. laryngeal cancer) or diagnosed voice condition
* Known brain or brainstem cancer
* Known head and neck cancer
* Known neurological disorders (i.e. stroke)
* Singers
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls: We shall recruit 8 normal healthy subjects (Group 1). Inclusion criteria for healthy controls include age >18 to 65 years old, non-smokers and no history of chronic respiratory symptoms. Asthmatics: We shall recruit a total of 16 patients with asthma - 8 patients with mild asthma (Group 2) and 8 patients with severe asthma (Group 3). Mild asthma will be defined as patients with forced expiratory volume in 1 second (FEV1) >80% predicted. Severe asthma will be defined as patients with FEV1 50-60% predicted. Asthmatics will also have a forced expiratory ratio (FER) less than the lower limit of normal, indicating obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Vocal cord aperture measured using continuous laryngoscopy after hyperventilation in normal subjects and asthmatics | 6 years
  For each experiment, the subject will sit in a comfortable armchair and breathe though a rubber mouthpiece and turbine pneumotachometer (Oxycon Delta, Jaeger, Wurzburg, Germany). The airflow and volume signals and that from the carbon dioxide (CO2) analyser will be displayed on a monitor and recorded. Subjects will breath through the spirometer during endoscopy to record respiratory phase for later correlation with laryngeal recording.
  Laryngeal movement analysis - Image stills will be taken from the continuous laryngoscopy recording, at end inspiration and end expiration. Measurement of narrowing of the laryngeal structures in relative terms during one breathing cycle, which is independent of the distance between the laryngoscope and the glottis.

SECONDARY OUTCOMES:
Lung function indices after hyperventilation in normal and asthmatic patients. | 6 years
  Spirometry indices after hyperventilation. Baseline spirometry will be recorded. Forced vital capacity (FVC) and forced expiratory volume (FEV1) will be calculated. Both are measurements of volume of air expired after maximum inspiration, measured in litres.
Role of the extra-thoracic airway hyper-responsiveness measured using bronchial provocation test to identify asthma like symptoms. | 6 years
  Role of the extra-thoracic airway hyper-responsiveness to asthma like symptoms using Mannitol bronchial provocation testing
Vocal cord changes after anti-cholinergic inhalers and/or exercise. | 6 years
  Vocal cord changes after anti-cholinergic inhalers and/or exercise. Subjects will inhale 4 puffs of ipratropium bromide (20 mcg/actuation inhalation) or placebo using normal tidal breathing. Subjects will then be exercised on an ergometer (Cateye Ergociser) at 75% to 85% of their predicted maximal heart rate (maximal heart rate equals 220 minus subjects age) for 8 minutes while breathing dry air at 10oC. Laryngoscopy will be conducted in situ as detailed in Project 1.
  Exercise will be discontinued and PVCM will be assessed. Final lung function testing will be performed to assess the degree of respiratory obstruction produced.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Ruane, BSc, Principal Investigator — Monash Health and Monash University
Locations (1):
- Monash Medical Centre, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Though publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: All